CLINICAL TRIAL: NCT03487211
Title: Comparative Efficacy of Duloxetine vs Escitalopram in Patients With Fibromyalgia
Acronym: CORTEX
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Responsible Party: Principal Investigator, DR. MOHAMMAD ALI ARIF, Assistant Professor of Medicine, Shaheed Zulfiqar Ali Bhutto Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShaheedZABMU
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia treatment; Duloxetine; Escitalopram
MeSH Terms: conditions — Fibromyalgia | interventions — Duloxetine Hydrochloride; Escitalopram

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant
Masking Description: Patients shall be provided medication with numeric labels
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Duloxetine Group (Active Comparator): Duloxetine 30mg once daily to be started for 1 week. Dose will then be titrated to 60mg once daily and the patients followed for a total of 12 weeks.
  Interventions: Drug: Duloxetine
- Escitalopram Group (Experimental): Escitalopram 10mg once daily to be started for 1 week. Dose will then be titrated to 20mg once daily and the patients followed for a total of 12 weeks.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Duloxetine — Duloxetine 30mg PO once daily for 1 week followed by an increase to 60mg PO once daily
  Other Names: DUPREX
  Arms: Duloxetine Group
Drug: Escitalopram — Escitalopram 10mg PO once daily for 1 week followed by an increase to 20mg PO once daily
  Other Names: EXAPRO
  Arms: Escitalopram Group

SUMMARY:
Duloxetine is FDA approved as pharmacological treatment for Fibromyalgia. The use of SSRIs has been endorsed by the 2013 Canadian guidelines. The data available for Escitalopram as a treatment modality for Fibromyalgia is limited, however small trials have demonstrated its efficacy. No head to head comparisons between escitalopram and duloxetine have been undertaken. We aim to conduct a single blind, randomized control trial to assess the comparative efficacy of duloxetine vs escitalopram in drug naive patients with newly diagnosed Fibromyalgia.

DETAILED DESCRIPTION:
180 drug naive patients with newly diagnosed fibromyalga according to the modified ACR 2016 criteria shall be enrolled by consecutive sampling after taking written informed consent. Baseline severity of fibromyalgia shall be assessed via the Revised Fibromyalgia Impact Questionnaire (FIQ-R). They shall be randomized via cluster randomization into two groups. The first group shall receive Duloxetine 30mg, will be increased to 60mg after one week. The second group shall receive Escitalopram 10mg to be increased to 20mg after one week. Patients shall be followed at 0,2,4,8 and 12 weeks. At each visit, any subjective change in symptoms shall be noted and the FIQ-R shall be re administered. At the end of the trial, the overall change in the FIQ-R from baseline shall be assessed and the difference between both groups will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Drug Naive patients
* Newly diagnosed with FIbromyalgia according to Modified ACR 2016 criteria

Exclusion Criteria:

* Concomitant depression/bipolar disorder or any other documented psychiatric illness
* Autoimmune disorders (SLE, RA)
* Peripheral Neuropathic pain due to any cause
* Uncontrolled hypertension
* Impaired renal or hepatic functions (on Lab assay)
* Chronic infections (e.g.Tuberculosis)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Reduction in FIQ-R (Revised Fibromyalgia Impact Questionnaire) from baseline | 4,8 and 12 weeks
  Percentage decrease in FIQ-R from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad A Arif, MRCP, FRCP, Principal Investigator — Shaheed Zulfiqar Ali Bhutto Medical University
Locations (1):
- Pakistan Institute of Medical Sciences, Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bennett RM, Bushmakin AG, Cappelleri JC, Zlateva G, Sadosky AB. Minimal clinically important difference in the fibromyalgia impact questionnaire. J Rheumatol. 2009 Jun;36(6):1304-11. doi: 10.3899/jrheum.081090. Epub 2009 Apr 15. PMID 19369473
- [Result] Wright CL, Mist SD, Ross RL, Jones KD. Duloxetine for the treatment of fibromyalgia. Expert Rev Clin Immunol. 2010 Sep;6(5):745-56. doi: 10.1586/eci.10.64. PMID 20828282
- [Result] Smith HS, Bracken D, Smith JM. Pharmacotherapy for fibromyalgia. Front Pharmacol. 2011 Mar 31;2:17. doi: 10.3389/fphar.2011.00017. eCollection 2011. PMID 21772818